CLINICAL TRIAL: NCT03748472
Title: The Effects of Bolus Feeding as Compared to Continuous Gavage Feeding on the Oxygenation Instability During Feeds Among Premature Infants
Brief Title: The Effect of Feeding Length on the Oxygenation Instability Among Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Liron Borenstein MD, Neonatologist, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Feeding length and oxygenation
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Premature Infant; Respiratory Disease
MeSH Terms: conditions — Premature Birth; Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus feeding (Experimental)
  Interventions: Procedure: Bolus feeding
- continuous gavage feeding (Experimental)
  Interventions: Procedure: Continuous gavage feeding

INTERVENTIONS:
Procedure: Continuous gavage feeding — Each subject will serve as his or her own control. In this arm infants will receive their feed over 2 hours and the next feed will be given over 30 min and then over 2 hours again.
  Arms: continuous gavage feeding
Procedure: Bolus feeding — Each subject will serve as his or her own control. In this arm infants will receive their feed over 30 min and the next feed will be given over 2 hours and then over 30 minutes again.
  Arms: Bolus feeding

SUMMARY:
SpO2 instability is in the nature of premature infants. Hypoxic episodes occur spontaneously in many of these infants, especially after the first week of life. Different interventions have been shown to influence the incidence of hypoxemic episodes in premature infants. Premature infants are fed via an NG/OG tube. Feeding length might influence the oxygenation instability among premature infants therefore the aim of this study is to evaluate the changes in oxygenation among preterm infants receiving respiratory support when are fed over 30 min vs over 2 hours, as documented by SpO2 histograms.

ELIGIBILITY:
Inclusion Criteria:

Premature Infants (GA<37weeks) on non-invasive respiratory support (CPAP, NIPPV, HFNC) Feeding>100 ml/kg/day

Exclusion Criteria:

Congenital anomalies e.g. gastroschesis, congenital diaphragmatic hernia, cyanotic heart disease.

Instability because of:

Acute lung pathology for example x-ray confirmed pneumonia, air leak Active culture proven sepsis Need for inotropic support for low blood pressure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Oxygenation instability | 9 hours (3 feeds)
  SPO2 histogram documents the oxygenation stability. we will record the histogram at the end of each period of time and compare it

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided